CLINICAL TRIAL: NCT01234012
Title: A Phase I Study of Therapeutic Cancer Vaccine IMF-001 in Patients With Malignancies Expressing NY-ESO-1
Brief Title: Study of IMF-001 in Patients With Malignancies Expressing NY-ESO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoFrontier, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMF001-PRT001
Record Dates: First submitted 2010-10-26; First posted 2010-11-04 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Solid Tumor
Keywords: melanoma; breast cancer; ovarian cancer; prostate cancer; esophageal cancer; uterine cancer; sarcoma; NY-ESO-1
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms; Uterine Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment: IMF-001 (Experimental): 100 or 200 mcg will be administered to patients subcutaneously every 2 weeks for 6 injections.
  Interventions: Biological: IMF-001

INTERVENTIONS:
Biological: IMF-001 — subcutaneous injection of fixed dose IMF-001 (100 or 200 mcg) every 2 weeks.

SUMMARY:
The purpose of this study is assess the safety of administering repeated doses of IMF-001, a vaccine, to patients with solid tumors that express NY-ESO-1 antigen. If the vaccine is therapeutically useful, a second goal is to establish the maximum therapeutic dose to treat patients with NY-ESO-1 positive cancers.

DETAILED DESCRIPTION:
NY-ESO-1 was isolated by serological analysis of recombinant cDNA expression libraries (SEREX), using tumor mRNA and autologous serum from an esophageal cancer patient. Reverse transcription-polymerase chain reaction (RT-PCR) analysis showed that NY-ESO-1 displayed the typical expression pattern of cancer testis antigens (CT antigens). NY-ESO-1 mRNA was expressed only in testis of normal tissues tested and in various types of cancer, including lung cancer, breast cancer, malignant melanoma and bladder cancer. Since testis is an immune privileged organ where HLA molecules are not expressed, these antigens can be considered tumor-specific.

IMF-001 is a CHP-NY-ESO-1 complex consisting of recombinant NY-ESO-1 protein and cholesteryl hydrophobized pullulan (CHP). CHP forms colloidally stable nanoparticles in water and complexes with substrate such as NY-ESO-1 protein.

It is well known that exogenous antigen proteins can induce specific CD4+ T cells but not specific CD8+ T cell. Dendritic cells pulsed with IMF-001 induced NY-ESO-1 specific CD8+ T cells in blood samples of 4 healthy volunteers. These data suggest that immunization of patients with IMF-001 can evoke not only specific CD4+ T cells responses but also specific CD8+ T cell response to NY-ESO-1 more effectively than NY-ESO-1 protein alone. Similar results for both cellular and humoral immunity in response to NY-ESO-1 protein were observed in previous clinical investigational studies with IMF-001.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven progressive or metastatic solid tumors expressing NY-ESO-1, who have failed standard treatment and have no other effective treatment available (solid tumors such as melanoma, breast cancer, ovarian cancer, prostate cancer, esophageal cancer, uterine cancer, and sarcoma frequently express NY-ESO-1). Patients with malignant melanoma stages IIb and III, or stage IV melanoma that has been completely resected, or with stage I and II uterine serous cancer, clear cell carcinoma, or carcinosarcoma with documented expression of NY-ESO-1 may also enroll as they have a 50% or greater chance of developing recurrent disease.
2. Documentation of tumor cells expressing NY-ESO-1 antigen as determined by immunohistochemistry.
3. Must have target lesion(s) measurable or non-measurable by RECIST version 1.1. Exceptions: Patients with stages IIb or III melanoma, or stage IV melanoma that has been completely resected, will have no target lesions measurable by RECIST version 1.1 but may enroll; patients with prostate cancer without measurable disease but with rising prostate specific antigen (PSA) levels may enroll; patients with resected stage I and II uterine serous cancer, clear cell carcinoma, and carcinosarcoma will have no target lesions measurable by RECIST but may enroll.
4. Has recovered from all acute adverse effects of prior therapy, with the exception of alopecia.
5. Laboratory values within the following limits:

   * Hemoglobin ≥ 8.0 g/dL
   * WBC count ≥ 2.0 x 10^9/L
   * ANC ≥ 1.0 x 10^9/L
   * Platelet count ≥ 75 x 10^9/L
   * Serum creatinine ≤ 1.5 mg/dL
   * AST & ALT ≤ 2.5 x ULN (≤ 5 x ULN if with hepatic metastases)
   * Serum total bilirubin ≤ 1.5 x ULN
6. Performance status of 0 or 1 (ECOG Scale).
7. Life expectancy ≥ 4 months.
8. Ages 18 years or over.
9. Patients with central nervous system metastases may be included if they are treated and stable for 2 months without the need for administration of steroids. Patients with unstable metastatic CNS disease are excluded.
10. A negative pregnancy test must be documented at the screening/baseline visit for women of childbearing potential. A female patient of childbearing potential, and a male patient with a female partner of childbearing potential, must be using at least one form of Investigator-approved contraception while on-study and for at least 1 month after their last administration of study therapy.
11. Able and willing to give written informed consent.

Exclusion Criteria:

1. Clinically significant heart disease (NYHA Class III or IV).
2. Serious active infection requiring antibiotics.
3. Bleeding disorders.
4. Unstable metastatic disease in the central nervous system.
5. Concomitant systemic treatment with corticosteroids. Topical steroids are permitted.
6. History of any severe or life-threatening hypersensitivity or allergic reaction.
7. Known HIV infection.
8. History of immunodeficiency disease or autoimmune disease, including scleroderma, Sjögren's syndrome, lupus erythematosus, idiopathic thrombocytopenic purpura (ITP), multiple sclerosis, or rheumatoid arthritis.
9. Has received anticancer chemotherapy, immunotherapy, radiotherapy or any other investigational agent within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to enrollment. Concomitant immunosuppressive therapy is not permitted. Adjuvant interferon alpha is not allowed for patients with stages IIb, III or IV melanoma. Prostate cancer patients with PSA only recurrence may have had previous androgen deprivation therapy, provided the 4 week washout period is observed.
10. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability of repeat doses. | Date of first dose until 30 days after off-study, or until resolution of related AEs

SECONDARY OUTCOMES:
Tumor response using RECIST 1.1 | Each cycle at weeks 7 and 11 (appx.)
  Scans will be performed each cycle after the 4th and 6th injections (approximately Weeks 7 and 11). Scans will be performed; or, for patients with prostate cancer, response will be based on PSA levels.
Humoral and cellular immune response as indication of IMF-001 biologic activity | Starting from first dose, samples taken within 72hrs of the 1st, 3rd, and 5th doses of each cycle until off-study
  Humoral response (NY-ESO-1 antibody titre) Cellular response (NY-ESO-1 specific CD4 and CD8 T-cells)
Optimal dose based on number of patients with adverse events at that dose | Date of first dose until 30 days after off-study, or until resolution of related AEs

CONTACTS AND LOCATIONS:
Overall Officials: DAIJU ICHIMARU, BS, Study Director — ImmunoFrontier, Inc.
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University (NYU) Cancer Center, New York, New York